CLINICAL TRIAL: NCT01784952
Title: Consumption of Whole Grains and Legumes Modulates the Genetic Effect of the APOA5 -1131C Variant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: WG_APOA5
Record Dates: First submitted 2013-02-03; First posted 2013-02-06 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Subjects With Mild Hypertriglyceridemia in Type 2 DM
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole grains and lequmes (Experimental)
  Interventions: Dietary Supplement: Dietary intervention
- refined rice (Placebo Comparator)
  Interventions: Dietary Supplement: Dietary intervention

INTERVENTIONS:
Dietary Supplement: Dietary intervention — The intervention program consisted of replacing of refined rice intake with 1/3 of legumes, 1/3 of barleys, and 1/3 of whole grains three times per day as a high carbohydrate source and increased vegetable intake to at least 6 units (30-70 g/unit) per day for sufficient dietary fiber intake. The subjects were recommended to drink no more than one alcoholic beverage drink (15 g alcohol) per day and were assigned physical activity consisting of a regular 30-min walk after dinner each day. Participants were also instructed to record their physical activity diary for 24 h every 4 weeks.

SUMMARY:
We examined whether a substitution of whole grains and legumes for refined rice in a high carbohydrate diet (about 65% of energy derived from carbohydrate) may modify the effect of this variant on changes in apolipoprotein A-V (apoA-V) and triglyceride concentrations.

DETAILED DESCRIPTION:
We genotyped the APOA5 -1131T>C in individuals with impaired fasting glucose (IFG) or newly diagnosed type 2 diabetes, who were randomly assigned to either a group ingesting whole grain and legume meals daily or a control group for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were in in impaired fasting glucose (IFG, 100≤ fasting glucose <126 mg/dL) and newly diagnosed type 2 diabetes (fasting glucose ≥126 mg/dL) were referred to the Department of Family Medicine or Internal Medicine. They were rechecked for their health and lipid profiles, and then those who satisfied the study criteria were recommended to participate in the dietary intervention program

Exclusion Criteria:

* Current and/or past history of cardiovascular disease including angina
* Liver or kidney dysfunction
* Thyroid or pituitary disease
* Unstable weight loss/gain (≥2 kg) over the previous 6months
* Pregnancy or lactation. Subjects who were taking medication were also excluded

Ages: 25 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Triglyceride | change from baseline in TG at 12 weeks

SECONDARY OUTCOMES:
Apolipoprotein A5 | Change from baseline in ApoA5 at 12 weeks

OTHER OUTCOMES:
Apolipoprotein A5 gene | ApoA5 -1131T>C polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph.D, Principal Investigator — Yonsei University
Locations (1):
- Yonsei university, Seoul, South Korea

REFERENCES:
- [Derived] Kang R, Kim M, Chae JS, Lee SH, Lee JH. Consumption of whole grains and legumes modulates the genetic effect of the APOA5 -1131C variant on changes in triglyceride and apolipoprotein A-V concentrations in patients with impaired fasting glucose or newly diagnosed type 2 diabetes. Trials. 2014 Apr 1;15:100. doi: 10.1186/1745-6215-15-100. PMID 24690159